CLINICAL TRIAL: NCT06886074
Title: Efficacy of Short-course Blinatumomab in Patients With Detectable Measurable Residual Disease With Philadelphia Chromosome-negative B-cell Acute Lymphoblastyc Leukemia
Brief Title: Efficacy of Short-course Blinatumomab for MRD Erradication in B-ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Head of Hematology, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE25-00007
Record Dates: First submitted 2025-03-03; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Acute Lymphoblastic Leukemia; Measurable Residual Disease (MRD)
Keywords: Blinatumomab; Measurable residual disease
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual

STUDY DESIGN:
Intervention Model Description: One arm, open-label, phase 2 study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blinatumomab arm (Experimental): Patients will receive 7 days of blinatumomab with a fixed dose of 175 mcg through out 7 days
  Interventions: Drug: Short course of blinatumomab

INTERVENTIONS:
Drug: Short course of blinatumomab — Patients will receive 175 mcg of blinatumomab trough out seven days in a 24-hours infusion.
  Blinatumomab therapy will be assigned 17.5 mcg per day for the first 2 days. Then blinatumomab 28 mcg per day for 5 days (completing 7 days). A single intravenous 20 mg dose of dexamethasone will be applied one hour before starting dose.

SUMMARY:
Detectable measurable residual disease (MRD) is the most important prognostic factor for B-cell acute lymphoblastic leukemia (B-ALL) for overall survival (OS) and disease-free survival (DFS). Patients who are MRD positive and have no access to novel immunotherapies should receive an allogeneic hematopoietic stem cell transplantation (HSCT). Blinatumomab is considered a standard of care (SOC) for this group of patients, however, the ideal treatment dose for MRD is unknown as doses were adjusted from the relapsed/refractory setting. Preliminary data suggest short cycles of blinatumomab can also be effective in states of lower disease burden prior to transplant. Thus, the investigators are performing a phase 2 trial assessing 7 days of blinatumomab as a bridge to HSCT

Primary endpoint is assessing the MRD response following a short-course blinatumomab infusion in patients with B-ALL with complete response (CR) and have detectable MRD disease who are candidates for HSCT. Secondary endpoints include incidence of adverse events, OS, DFS, percentage of patients who receive HSCT, incidence of cytokine release syndrome (CRS) and immune effector cell associated neurotoxicity syndrome (ICANS)

DETAILED DESCRIPTION:
During the proposed treatment, blinatumomab therapy will be assigned as follows:

Blinatumomab 17.5 mcg per day for 2 days, followed by blinatumomab 28 mcg per day for 5 days. Dexamethasone 20 mg will be applied one hour before starting dose.

The immunotherapy will be applied as a 24-hour continuous infusion. The scheduled appointments will be on the initial day of blinatumomab, when the patient will be discharged from hospital and evaluation will be performed on day 10 with bone marrow aspiration and MRD assessment trough next generation flow cytometry. The results will be given at the appointment on day 14, along with an assessment profile for HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Philadelphia chromosome-negative B-cell acute lymphoblastic leukemia
* MRD detectable in complete response (above the limit of quantification according to FCM)
* Performance status 0-2 on the ECOG scale
* No prior organ damage
* Having a potential related or unrelated donor

Exclusion Criteria:

* Performance status on the ECOG scale >2
* HCT-CI >3 points
* Patients who do not wish to participate in clinical study.
* Active central nervous system infiltration (CNS3)
* Active extramedullary disease
* Having previously received blinatumomab
* Absence of related or unrelated donors

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy to eradicate MRD in negative Philadelphia-chromosome B-cell acute lymphoblastic leukemia | 24 months
  Primary outcome is to determinate the efficacy of blinatumomab to eradicate MRD in a blood sample extracted by bone marrow aspiration and evaluated by next generation flow cytometry on the third day after blinatumomab completion (day 10 after initiation). MRD eradication will be defined as: undetectable (below limit of detection) disease through next generation flow cytometry.

SECONDARY OUTCOMES:
Overall survival | 24 months
  Survival time after enrollment
Disease free survival | 24 months
  Time from enrollment to relapse
Percentage of patients undergoing stem cell transplantation | 24 months
  Percentage of patients who undergo hematopoietic stem cell transplantation after enrollment
Incidence of adverse events | 24 months
  Incidence of hematologic (anemia, thrombocytopenia, leukopenia, neutropenia, lymphocytopenia) and non-hematologic (renal, hepatic, dermatologic, cardiovascular, infectious) adverse events after initiating blinatumomab therapy assessed by CTCAE V 5.0
Incidence of cytokine release syndrome | 24 months
  Incidence and grading of cytokine release syndrome after initiating blinatumomab through CTCAE V 5.0
Incidence of immune effector cell-associated neurotoxicity syndrome | 24 months
  Incidence and grading of immune effector cell-associated neurotoxicity syndrome after initiating blinatumomab assessed by ASTCT grading system.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Dr. Jose E. Gonzalez, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Yin J, Cai X, Qian B, Liu Y, Li D. Short-Course Blinatumomab Treatment as a Bridge to Further Salvage Therapy for Relapsed/Refractory B-Cell Acute Lymphoblastic Leukemia: A Retrospective Single-Center Study. Cancer Med. 2024 Dec;13(24):e70515. doi: 10.1002/cam4.70515. PMID 39692275